CLINICAL TRIAL: NCT02806115
Title: The Efficacy of Severe Whitening and Delayed Fading in Acetic Acid-enhanced Endoscopy for Diagnosing Gastric Intestinal Metaplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015SDU-QILU-G003
Record Dates: First submitted 2016-06-05; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Intestinal Metaplasia
MeSH Terms: interventions — Acetic Acid; Endoscopes

ARMS (1):
- acetic acid-enhanced endoscopy (Experimental): Acetic acid-enhanced endoscopy combines conventional endoscopy with the instillation of acetic acid.
  Interventions: Procedure: acetic acid-enhanced endoscopy; Drug: Acetic Acid; Device: endoscope

INTERVENTIONS:
Procedure: acetic acid-enhanced endoscopy — Acetic acid-enhanced endoscopy combines conventional endoscopy with the instillation of acetic acid.
Drug: Acetic Acid — The concentration of acetic acid used in this study is 1.5%.
Device: endoscope — This study using an EG-29-i10 endoscope (Pentax, Tokyo, Japan) and an EPK-i7010 processor (Pentax, Tokyo, Japan).

SUMMARY:
Investigators found that the degree and the duration of aceto-whitening differed between gastric intestinal metaplasia(GIM) and the surrounding normal mucosa: the area of GIM showed a severe degree of aceto whiteness and the whitening continued longer than the surrounding normal mucosa, which investigators called "severe whitening" and "delayed fading", and investigators realized that GIM could possibly be diagnosed by using these differences.The aim of this prospective study was to investigate the efficacy of "severe whitening" and "delayed fading" for diagnosing GIM.

ELIGIBILITY:
Inclusion Criteria:

* long-lasting upper gastrointestinal symptoms (>15 years)
* atrophic gastritis or GIM identified at surveillance endoscopy

Exclusion Criteria:

* presence of advanced adenocarcinoma in the stomach
* presence of acute gastrointestinal bleeding
* presence of coagulopathy, uncontrolled impaired renal or liver disease
* presence of pregnancy or lactation
* presence of allergy to acetic acid
* age younger than 18 years or older than 80 years
* inability to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
accuracy of "severe whitening" for diagnosing gastric intestinal metaplasia | 6 months
accuracy of "delayed fading" for diagnosing gastric intestinal metaplasia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China